CLINICAL TRIAL: NCT06086847
Title: Effects of Progressive Resistance Training on Physical State Energy and Fatigue During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0530
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Pregnancy Related
Keywords: Energy state; Fatigue; Pregnancy; Muscle stretching exercises
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm up Exercise + stretching Exercise + progressive resistance exercises (Experimental): * Group A (Experimental Group):
  * Warm up Exercise + stretching Exercise (upper and lower extremity) + progressive resistance exercises Warm up Exercise (for 5 min) Stretching (upper and lower extremity)
    3. Progressive Resistance exercises:
    1. Leg press :( dual leg press): Leg press target the
       "Quadriceps" or quads .but they also work your "Hamstrings".
    2. Leg curls (dual leg curls):
  Leg curls Target the "hamstrings" and "Calf" muscles Leg Extension
  The Muscles worked:
  1. Rectus femoris
  2. Vastus lateralis
  3. Vastus medialis
  4. Vastus intermedius
  4. Arm lat pull (dual arm lat pull):
  Back extension (lumber extension):
  Interventions: Other: progressive resistant exercises
- warm up exercise + Stretching exercises (Active Comparator): Warm up exercise (for 5 min)
  Stretching exercises (upper and lower extremity
  Interventions: Other: progressive resistant exercises

INTERVENTIONS:
Other: progressive resistant exercises — Group A (Experimental Group):
  • Warm up Exercise + stretching Exercise (upper and lower extremity) + progressive resistance exercises Warm up Exercise (for 5 min) Stretching (upper and lower extremity)
  3. Progressive Resistance exercises:
  1. Leg press :( dual leg press): Leg press target the
     "Quadriceps" or quads .but they also work your "Hamstrings".
  2. Leg curls (dual leg curls):
  Leg curls Target the "hamstrings" and "Calf" muscles Leg Extension
  The Muscles worked:
  1. Rectus femoris
  2. Vastus lateralis
  3. Vastus medialis
  4. Vastus intermedius
  4. Arm lat pull (dual arm lat pull):
  Back extension (lumber extension):

SUMMARY:
The purpose of this study is to compare the effects of progressive resistance training on physical state energy and fatigue during pregnancy. This study was a randomized controlled trial used to find the effects of progressive resistance training on physical state energy and fatigue during pregnancy. The data was collected from Sheikh Zaid Hospital via Visual analogue scale-fatigue, Numeric pain rating scale and Short form health survey-36. Sample size of 30 females was taken in 15 each group.

DETAILED DESCRIPTION:
According to the findings of a study on physical activity during pregnancy in 2021, obese women, who exercise less than ladies of normal body weight may gain from gradually increasing their amount of exercise to reduce the amount of weight gain associated with pregnancy. Exercise during pregnancy was consistently associated positively with sob-R among the women in both categories, which denotes that it may have an impact on the control of lepton activity and pregnancy-induced insulin resistance. Overall, our research suggests that obese women, who are lepton-resistant and at pregnant women at high risk of gestational diabetes, fast weight gain, and increased fetal adiposity should receive advice and supportive services to raise their activity level, with an emphasis on the fact that even slight improvements in action can be good for both child and maternal health.

ELIGIBILITY:
Inclusion Criteria:

* Female with age of 20 to 40 years
* Between 20-25 weeks of gestation.
* Healthy individual
* Pregnant females who are easily fatigued during activities of daily living.

Exclusion Criteria:

* • Those who reported regular resistance training exercises

  * Complicated pregnancy
  * Low pre-pregnancy body weight
  * Anemia
  * Diabetes
  * Psychiatric disorder
  * Orthopedic and cardiovascular limitation

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy only occurs in females.
Enrollment: 28 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Short Form Health survey (SF-36) | 9 WEEKS
  Eight dimensions of health-related quality of life are measured using the 36-item Short Form Health Survey (SF-36). 36 items make up the questionnaire, which assesses physical functioning, role restrictions brought on by physical health, physiological discomfort, overall health status, vitality, social functioning, role limitations brought on by emotional issues, and mental health. A substantial body of research supports the reliability of the SF-36 measurements
Numeric Pain Rating Scale(NPRS) | 9 WEEKS
  The patient's level of pain is recorded by the NPRS (intensity of pain). Patients are asked to rate their current degree of pain on an 11-point scale with 0-3 representing mild pain, 4-6 representing moderate pain, and 7- 10 representing severe pain (Severe pain). Horizontal bars or lines are the standard format.
Visual Analogue Scale-Fatigue(VAS-F) | 9 WEEKS
  The scale has 18 components that are all related to one's perception of exhaustion. Each question asks respondents to place a "X" along a visual analogue line that runs between two extremes, such as "not at all fatigued" and "very tired," to indicate how they are feeling right now. Scores range from 0 to 100 due to the length of each line being 100 mm. Moreover, the instrument has two subscales: weariness (items 1-5, 11- 18), and energy (items 6-10)

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Taufiq, PPDPT, Principal Investigator — Riphah International University, Senior Lecturer
Locations (1):
- Family Health Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No